CLINICAL TRIAL: NCT01423253
Title: A 12-Week, Open-Label Extension Study For the Treatment of Major Depressive Disorder With Mixed Features
Brief Title: Major Depressive Disorder With Mixed Features - Extension
Acronym: RESOLVE3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D1050306
Record Dates: First submitted 2011-08-23; First posted 2011-08-25 (Estimated); Results first posted 2015-10-14 (Estimated); Last update posted 2016-04-08 (Estimated); Status verified 2016-03

CONDITIONS: Major Depressive Disorder
Keywords: Depression; Lurasidone; Latuda
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Lurasidone Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lurasidone 20, 40, 60 mg (Experimental): Lurasidone 20, 40, or 60 mg/day flexibly dosed
  Interventions: Drug: Lurasidone

INTERVENTIONS:
Drug: Lurasidone — Lurasidone 20, 40, or 60 mg/day, orally, once daily (QD) in the evening, with a meal or within 30 minutes after eating, flexibly dosed
  Other Names: Latuda

SUMMARY:
Lurasidone HCl is a compound that is a candidate for the treatment of major depressive with mixed features.This clinical study is designed to test how well Lurasidone works to treat major depressive disorder with mixed features over time.

ELIGIBILITY:
Inclusion Criteria:

Subject provides written informed consent and is willing and able to comply with the protocol in the opinion of the Investigator.

Subject has completed 6 weeks of treatment in Study D1050304 (NCT#01421134) or Study D1050305 (NCT#01423240).

Subject is judged by the Investigator to be suitable for participation in a 12-week clinical trial involving open-label lurasidone treatment and is able to comply with the protocol in the opinion of the Investigator.

Exclusion Criteria:

Subject answers "yes" to "Suicidal Ideation" Item 4 or 5 on the C-SSRS (at time of evaluation) at baseline (Day 43 in Study D1050304 or D1050305).

Subject is considered by the Investigator to be at imminent risk of suicide or injury to self, others, or property.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2011-09; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, MD, Study Director — Sumitomo Pharma America, Inc.
Locations (17):
- United States (17):
  - Birmingham Psychiatry Pharmaceutical Studies, Inc, Birmingham, Alabama
  - Synergy Clinical Research Center, Escondido, California
  - Collaborative Neuro Science Network, Inc., Garden Grove, California
  - Stanford -VA Palo Alto Health Care System, Palo Alto, California
  - Artemis Institute for Clinical Research, San Diego, California
  - Florida Clinical Research Center, LLC, Sarasota, Florida
  - Massachusetts General Hospital - Center for Anxiety and Traumatic Stress Disorders, Boston, Massachusetts
  - St. Charles Psychiatric Associates/Midwest Research Group, Saint Charles, Missouri
  - Village Clinical Research Inc., New York, New York
  - Finger Lakes Clinical Research, Rochester, New York
  - Behavioral Medical Research of Staten Island, Staten Island, New York
  - Psychiatry and Behavioral Sciences, Duke, Durham, North Carolina
  - Midwest Clinical Research Center, Dayton, Ohio
  - CRI Worldwide - Kirkbride, Philadelphia, Pennsylvania
  - FutureSearch Trials of Dallas, LP, Dallas, Texas
  - Dept. of Psychiatry, UT Southwestern Medical Center, Dallas, Texas
  - Grayline Clinical Drug Trials, Wichita Falls, Texas

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lurasidone 20, 40, 60 mg
Started | 48
Completed | 39
Not Completed | 9
Not completed — Adverse Event | 2
Not completed — Lack of Efficacy | 2
Not completed — Lost to Follow-up | 1
Not completed — Protocol Violation | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Population: Safety population
Arm/Group | Lurasidone 20, 40, 60 mg
Number analyzed (Participants) | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 45
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42.5 (13.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36
  Male | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 21
  White | 24
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 48

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Treatment Emergent Adverse Events (TEAEs)
Description: Percentage of subjects with treatment emergent adverse events (TEAEs)
Time Frame: 12 Weeks
Population: Safety population
Measure: Number; unit: percentage of subjects
Arm/Group | Lurasidone 20, 40, 60 mg
Number analyzed (Participants) | 48
percentage of subjects | 66.7

2. Secondary Outcome: Mean Change From Baseline to Week 12 (LOCF) in MADRS Total Scores
Description: Mean change from baseline to week 12 (LOCF) in Montgomery-Asberg Depression Rating Scale (MADRS) total scores The MADRS is a clinician-rated assessment of the subject's level of depression and consists of 10 items. Each item is rated on a Likert scale, from 0="Normal" to 6="Most Severe". The MADRS total score is calculated as the sum of the ten items and ranges from 0 to 60. Higher scores are associated with greater severity.
Time Frame: Baseline to12 Weeks
Population: Safety population - only 47 subjects had the MADRS assessment at Week 12 (LOCF).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lurasidone 20, 40, 60 mg
Number analyzed (Participants) | 47
units on a scale | -5.9 (12.94)

3. Primary Outcome: Percentage of Subjects With Treatment Emergent Serious Adverse Events (TESAEs)
Description: Percentage of subjects with Treatment Emergent Serious Adverse Events (TESAEs)
Time Frame: 12 Weeks
Population: Safety Population
Measure: Number; unit: percentage of subjects
Arm/Group | Lurasidone 20, 40, 60 mg
Number analyzed (Participants) | 48
percentage of subjects | 0

4. Primary Outcome: Percentage of Subjects Who Discontinued Due to Treatment Emergent Adverse Events (TEAEs)
Description: Percentage of subjects who discontinued due to Treatment Emergent Adverse Events (TEAEs)
Time Frame: 12 Weeks
Population: Safety Population
Measure: Number; unit: percentage of subjects
Arm/Group | Lurasidone 20, 40, 60 mg
Number analyzed (Participants) | 48
percentage of subjects | 4.2

5. Secondary Outcome: Change From Baseline to Week 12 (LOCF) in CGI-S Score
Description: The Clinical Global Impression - Severity of illness (CGI-S) score is a single value, clinician-rated assessment of illness severity and ranges from 1= 'Normal, not at all ill' to 7= 'Among the most extremely ill patients'. A higher score is associated with greater illness severity.
Time Frame: baseline to week 12
Population: Safety population - 1 subject did not have the CGI-S assessment at week 12 (LOCF)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lurasidone 20, 40, 60 mg
Number analyzed (Participants) | 47
units on a scale | -0.47 (1.442)

6. Secondary Outcome: Change From Baseline to Week 12 (LOCF) in the YMRS Total Score
Description: The Young Mania Rating Scale (YMRS) is an 11-item instrument used to assess the severity of mania. Seven items are rated on a 5-point scale, ranging from 0 to 4, and four items are rated on a 9-point scale, ranging from 0 to 8. The YMRS total score is calculated as the sum of the 11 items and ranges from 0 to 60. Higher scores are associated with greater severity of mania.
Time Frame: Baseline to week 12
Population: Safety population - 2 subject did not have YMRS assessment at week 12 (LOCF)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lurasidone 20, 40, 60 mg
Number analyzed (Participants) | 46
units on a scale | -1.5 (6.17)

7. Secondary Outcome: Change From Baseline to Week 12 (LOCF) in the HAM-A Total Score
Description: The Hamilton Rating Scale for Anxiety (HAM-A) is used to quantify the severity of anxiety symptomatology and consists of 14 items. Each item is rated on a 5-point scale, ranging from 0 (not present) to 4 (severe/disabling). The HAM-A total score is calculated as the sum of the 14 individual items and ranges from 0 to 56. Higher scores are associated with greater degree of anxiety.
Time Frame: Baseline to week 12
Population: Safety Population - 4 subjects did not have the HAM-A assessment at week 12 (LOCF)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lurasidone 20, 40, 60 mg
Number analyzed (Participants) | 44
units on a scale | -1.5 (6.48)

8. Secondary Outcome: Change From Baseline to Week 12 (LOCF) in the SDS Total Score
Description: The Sheehan Disability Scale (SDS) is a composite of three self-rated items designed to measure the extent to which three major sectors (work/school, social life/leisure, and family life/home responsibility) in the patient's life are impaired by depressive symptoms. These three items are responded to on a visual analogue scale (VAS) ranging through 0 (no impairment), 1-3 (mild), 4-6 (moderate), 7-9 (marked) and 10 (extreme) disability. The SDS total score is calculated as the sum of the three items and ranges from 0 (unimpaired) to 30 (highly impaired).
Time Frame: Baseline to week 12
Population: Safety Population - 12 subjects did not have the SDS total score at week 12 (LOCF)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lurasidone 20, 40, 60 mg
Number analyzed (Participants) | 36
units on a scale | -3.6 (9.95)

ADVERSE EVENTS:
Time Frame: 12 Weeks
Arm/Group | Lurasidone 20, 40, 60 mg
Serious Adverse Events (participants affected / at risk) | 0/48
Other Adverse Events (participants affected / at risk) | 16/48
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lurasidone 20, 40, 60 mg (N=48)
Diarrhoea (Gastrointestinal disorders) | 4 (4)
Nausea (Gastrointestinal disorders) | 3 (3)
Fatigue (General disorders) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 4 (4)
Akathisia (Nervous system disorders) | 5 (6)
Headache (Nervous system disorders) | 3 (4)
Sedation (Nervous system disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There IS agreement between Principal Investigator and Sponsor that restricts PI's rights to discuss or publish trial results after trial is completed.

In addition to the <60-180 day restriction above, since this is a multicenter study, 1st publication of study results shall be made with other participating study sites as a multicenter publication provided, if a multicenter publication is not forthcoming within 24 months post completion of study at all sites, PI shall be free to publish.